CLINICAL TRIAL: NCT04763850
Title: Effects of Real-time Feedback During Decline Walking on Kinematic and Kinetic Gait Parameters (Up & Down)
Brief Title: Effects of Real-time Feedback During Decline Walking on Kinematic and Kinetic Gait Parameters in a Healthy Population
Acronym: Up_and_Down
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Widhalm (Other)
Responsible Party: Sponsor-Investigator, Klaus Widhalm, Academic Staff, FH Campus Wien, University of Applied Sciences
Organization: FH Campus Wien, University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: project2010559
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Real-time feedback; Decline walking; Leg alignment; Kinematic; Kinetic; Treadmill

STUDY DESIGN:
Intervention Model Description: The study is set up as cross-sectional observation of gait under four conditions, which follows a randomized sequence in order to avoid carry over effects. Chronologically, the assessments will start with the tertiary observation, investigating agreements between declined/inclined ramp and treadmill walking. Thereafter, three out of four conditions (self-paced walking, self-paced walking with internal focus of attention, and self-paced walking with real-time feedback) are tested under block randomization of their six possible permutations . With three conditions (n=3), this represents the smallest number of permutations, equaling a Williams design, where each condition precedes each other condition equally often and each treatment occurs equally frequently at each position. The fourth corresponding condition (speed-matched walking) is exempted from the sequence randomization and always follows after self-paced walking with real-time feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking decline (Experimental): Walking decline on an instrumented treadmill under 3 different conditions
  Interventions: Other: Decline Walking with real-time Feedback

INTERVENTIONS:
Other: Decline Walking with real-time Feedback — Participants are walking decline with self-paced speed on an instrumented treadmill with virtual reality projection under three conditions: without instruction, with instruction for an internal focus of attention and with real-time feedback of their frontal knee alignment
  Other Names: Decline Walking with increased internal focus of attention; Decline Walking

SUMMARY:
Control of the dynamic functional leg alignment (dFLA) and biomechanical load are important joint related aspects regarding the development of osteoarthritis (OA). Research on level walking with feedback on load related parameters provided innovative treatment possibilities. Concerning walking on sloped surfaces, fundamental biomechanical knowledge exists. However, deeper insights into the control of the dFLA during decline walking, and the usefulness of real-time feedback are missing.

This study is set up as cross-sectional observation of gait under four conditions, which follows a randomized sequence in order to avoid carry over effects. Thirty (30) participants aged between 18 and 35 years will be included. They will complete a three-dimensional gait analysis on a 5-m ramp with 10° inclination. Afterwards they will be observed under four different conditions a) self-paced walking b) self-paced walking with internal focus of attention, c) self-paced walking with real-time feedback, and d) condition c speed-matched walking, on a 10° declined split belt treadmill. The primary outcome parameter will be the frontal knee range of motion (fKROM). Secondary outcomes include the ground reaction force loading rate, spatial-temporal parameters, sagittal frontal and transversal kinematics, and kinetics for the lower extremities.

The findings should improve the understanding of effects of real-time feedback on the control of the dFLA and lower limb loading. Results will be published in a peer-review journal.

ELIGIBILITY:
Inclusion Criteria:

1. age from 18-35 years
2. body mass index from 18.5 to 29.99 kg/m²
3. no chronical joint diseases and/or OA surgery
4. no neuro-motor diseases

Exclusion Criteria:

1. non-physiological and non-symmetrical gait patterns
2. severe outliers (more than two standard deviations)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
frontal knee range of motion during stance phase | during intervention
  frontal knee range of motion [degree]

SECONDARY OUTCOMES:
ground reaction force loading ratio | during intervention
  ground reaction force loading ratio [newton per second]

OTHER OUTCOMES:
3D kinematics of the lower limb | during intervention
  joint angles [degree]
3D kinetics of the lower limb | during intervention
  external joint moments [newtonmetre per kilogram bodyweight] frontal knee moment impulses [newtonmeter per kilogram bodyweight per second]

CONTACTS AND LOCATIONS:
Locations (1):
- FH Campus Wien, University of Applied Sciences, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
A manuscript will be submitted to a journal with peer review process aiming for an open access publication. Coded raw data will be made available upon request and for non-commercial purposes after publication of the results.

REFERENCES:
- [Derived] Widhalm K, Durstberger S, Putz P. Effects of visual real-time feedback during decline walking on gait parameters: a crossover randomized trial. BMC Musculoskelet Disord. 2025 Dec 23. doi: 10.1186/s12891-025-09437-7. Online ahead of print. PMID 41430600
- [Derived] Widhalm K, Durstberger S, Putz P. Effects of real-time feedback during decline walking on kinematic and kinetic gait parameters in a healthy population: study protocol for a randomized trial - up and down. Trials. 2021 Jul 22;22(1):477. doi: 10.1186/s13063-021-05422-2. PMID 34294137

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT04763850/Prot_SAP_000.pdf